CLINICAL TRIAL: NCT00744731
Title: The Open Label Extension Portion of the Study Entitled A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter Study to Evaluate the Efficacy, Safety, and Tolerability of Carisbamate as Adjunctive Therapy in Subjects With Partial Onset Seizures.
Brief Title: An Open-Label Extension Study of the Safety and Tolerability of Carisbamate as Add-On Therapy in Patients With Partial Onset Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SK Life Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 333369EPY3014; CARISEPY3014
Record Dates: First submitted 2008-08-29; First posted 2008-09-01 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Epilepsy, Partial, Motor; Epilepsy, Complex Partial; Epilepsy, Simple Partial; Focal Motor Epilepsy
Keywords: Partial-onset Seizures; Simple Partial Seizures; Complex Partial Seizures
MeSH Terms: conditions — Epilepsy, Partial, Motor; Epilepsy, Complex Partial; Epilepsies, Partial; Seizures | interventions — S-2-O-carbamoyl-1-o-chlorophenyl-ethanol

ARMS (2):
- 001 (Experimental): placebo placebo for 1 week
  Interventions: Drug: placebo
- 002 (Experimental): carisbamate 400 mg/day to 1,200 mg per day
  Interventions: Drug: carisbamate

INTERVENTIONS:
Drug: placebo — placebo for 1 week
  Arms: 001
Drug: carisbamate — 400 mg/day to 1,200 mg per day
  Arms: 002

SUMMARY:
The purpose of this study is to obtain long-term safety and tolerability information on carisbamate as add-on therapy for the treatment of partial onset seizures in patients with epilepsy. Seizure counts will be obtained to measure the rate of seizures for each patient during the study.

DETAILED DESCRIPTION:
CARISEPY3014 is the open-label extension study that follows the double-blind study CARISEPY3013 (NCT00740623). In an open label study such as CARISEPY3014, both the physician and the patient know the name of the assigned study medication. In a double blind study such as CARISEPY-3013, neither the physician nor the patient knows the name of the assigned study medication. Patients who complete the 14-week double-blind treatment phase of study CARISEPY3013 will be eligible to enter the open-label extension study during which patients will transition through a 1-week blinded period to open-label carisbamate. There will be a 1 week blinded transition during which patients will take blinded study medication; after this, patients will then take unblinded, open-label study medication. Safety assessments include the monitoring of the frequency, severity, and timing of adverse events, clinical laboratory test results, 12-lead electrocardiogram (ECG) recordings, vital signs measurements, physical and neurologic examinations, the Physician Withdrawal Checklist for symptoms of withdrawal for those patients who taper and/or discontinue study drug, and pregnancy tests for females of childbearing potential. Seizure counts will be obtained at every visit. The Quality of Life in Epilepsy-31 Patient Inventory questionnaire will be administered once during the study. A Medical Resource utilization questionnaire will be used to obtain cost-effectiveness information on carisbamate and will be administered twice during the study. There is no statistical testing hypothesis for this study. Carisbamate tablets taken twice daily in 2 equally divided doses, with or without food, and taken with noncarbonated water. During the first week on study, patients will take blinded transition study medication and thereafter will take a target dosage of 800 mg/day of unblinded, open-label study medication. The dosage of study medication will range from 400 to 1,200 mg/day. Patients will receive treatment for 1 year with the potential to receive treatment longer.

ELIGIBILITY:
Inclusion Criteria:

* Must have completed the 14-week double-blind treatment phase of study CARISEPY3013
* must be willing/able to follow the restrictions and prohibitions of the protocol
* must be able to complete the patient diaries correctly (patients or legally acceptable representatives)
* must sign an informed consent form indicating agreement to participate in the study (patients or legally acceptable representatives)
* adolescents capable of understanding the nature of the study must provide assent to participate in the study

Exclusion Criteria:

* Patients who have not completed the 14-week double-blind treatment phase of study CARISEPY3013.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 403 (Actual)
Dates: Start 2009-01; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Safety will be evaluated by the monitoring of the frequency, severity, and timing of adverse events, clinical laboratory test results, 12-lead electrocardiogram (ECG) recordings, vital signs measurements, physical and neurologic examinations | after a stable dose of Carisbamate is achieved, study visits to assess safety will be every three months for the duration of the subject's participation; subjects will also maintain a seizure count diary

SECONDARY OUTCOMES:
To evaluate the impact of carisbamate on subject functioning and well being using the QOLIE-31 Patient Inventory (as exploratory). Administered at month 3 and end of study. | after a stable dose of Carisbamate is achieved, study visits to assess safety will be every three months for the duration of the subject's participation; subjects will also maintain a seizure count diary

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.